CLINICAL TRIAL: NCT05789927
Title: Environmental Mycobiota: In-depth Characterisation and Determinants Involved in Asthma Emission
Acronym: MyCADO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/30
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Asthma
Keywords: mycobiota; Asthma; Environment
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — lung exacerbations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who received antibiotic prophylaxis: Severe "T2-High" asthmatics treated with biotherapy
  Interventions: Procedure: Assessment of the microbial exposome

INTERVENTIONS:
Procedure: Assessment of the microbial exposome — The assessment of the microbial exposome will be carried out by the deployment of 4 dust collectors (1 per season) at the patient's home. The evaluation of the endogenous myco-microbiome will be carried out by analyzing patient sputum obtained during follow-up visits or during routine care in the event of an exacerbation.

SUMMARY:
The analysis of the exposome of severe asthmatic patients and its correlation with the response profile to biotherapies used in the treatment of severe asthma and/or the frequency of exacerbations, could make it possible to identify individual and environmental components influencing the evolution of the asthmatic pathology and/or response to treatment. An interventional approach could thus be developed, taking into account in particular the determinants of indoor air quality as well as the obstacles to the implementation of current recommendations for the prevention of exacerbations.

The patient will thus be returned to the center and considered as a main actor in his clinical history by offering him the most suitable intervention possible, according to the evaluation of his exposome, in order to ultimately reduce the morbidity and mortality linked to exacerbations.

This interventional approach could then be validated on a larger scale in a national multicenter study involving a larger number of patients.

DETAILED DESCRIPTION:
Nowadays, 5 to 10% of the population of developed countries suffer from asthma, whose morbidity and mortality represent approximately 1% in years of life lost. Within this asthmatic population, there is a subgroup of patients with severe asthma (10% of total asthmatics). These severe asthma patients have a high risk of complications and exacerbations, poor quality of life, and increased mortality and morbidity. Moreover, these severe asthmatics represent 50% of the total health care costs associated with asthma. Among the formidable complications of severe asthma, exacerbations are still responsible for 900 deaths per year in France, while most of them are considered avoidable.

Severe asthma is currently described as a heterogeneous disease composed of multiple phenotypes, themselves linked to different pathophysiological mechanisms that define theendotypes. Phenotypic and endotypic characterization is important for the management of severe asthma, as recent therapeutic developments now make it possible to specifically target certain endotypes.In effect,in recent years, the development of new treatments using monoclonal antibodies (biotherapies) has improved the management of severe asthmatic patients with the "T2-High" phenotype, with a reduction in the frequency of exacerbations. However, the response to these new biotherapies is heterogeneous with super-responder patients (absence of exacerbations), partial responder patients (decrease but persistence of exacerbations) and non-responder patients (no effect on exacerbations).

Severe asthma, the diversity of phenotypes/endotypes observed, the frequency of exacerbations and the response to treatment, result from a combination of genetic and environmental factors. The exposome, which designates all of the exposures to external and environmental factors that a human undergoes from his development in utero until death, could therefore play a key role in the evolution of severe asthmatic pathology. Among these components of the exposome, the team find in particular microbial exposure (or environmental micro-mycobiota), including the omnipresent fungal spores in the air everybody breathe. Thus, in line with the hygienist hypothesis, recent studies have shown that environmental microbial exposures during early childhood, significantly reduced the incidence of respiratory disease in children with genetic susceptibility at chromosome 17q21. Additionally, chronic exposure to a microbial environment, particularly the fungal indoor environment, is associated with a wide range of adverse health effects, including asthma, and may influence its severity. More recently, severe asthma has also been associated with pulmonary microbial dysbiosis that would activate the inflammasome and other mediated pathways. However, the exposome is one of the factors that can influence this pulmonary microbial dysbiosis. particularly the fungal indoor environment, is associated with a wide range of adverse health effects, including asthma, and may influence its severity. More recently, severe asthma has also been associated with pulmonary microbial dysbiosis that would activate the inflammasome and other mediated pathways. However, the exposome is one of the factors that can influence this pulmonary microbial dysbiosis. particularly the fungal indoor environment, is associated with a wide range of adverse health effects, including asthma, and may influence its severity. More recently, severe asthma has also been associated with pulmonary microbial dysbiosis that would activate the inflammasome and other mediated pathways. However, the exposome is one of the factors that can influence this pulmonary microbial dysbiosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old,
* Patient with severe "T2-High" asthmatics,
* Treated with biotherapy for more than a year
* Regularly monitored at the University Hospitals of Bordeaux and Toulouse.

Exclusion Criteria:

* Severe asthmatic patients who have been treated with biotherapy for less than a year
* Severe asthmatic patients who have not been treated,
* Not Severe asthmatic patients
* Patient who are not regularly monitored at the Bordeaux and/or Toulouse University Hospitals
* Patients under the protection of justice, under guardianship, under curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion of patients will be done prospectively among patients > 18 years old, severe "T2-High" asthmatics treated with biotherapy for more than a year and regularly monitored at the University Hospitals of Bordeaux and Toulouse.The monitoring of the asthmatic pathology must also have been well carried out the year preceding inclusion in MyCADO, with in particular the evaluation of the initial response to biotherapy and the number of exacerbations that occurred during this year.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-04-17 (Estimated); Study Completion 2025-04-17 (Estimated)

PRIMARY OUTCOMES:
identify differences in bacterial and fungal of the microbial exposome | Month 3
  demonstration of an association between the components of the microbial exposome over an entire year and the response profile to biotherapies used in severe asthma (super-responder vs partial responders), evaluated according to Upham's criteria.
identify differences in bacterial and fungal of the microbial exposome | Month 6
  demonstration of an association between the components of the microbial exposome over an entire year and the response profile to biotherapies used in severe asthma (super-responder vs partial responders), evaluated according to Upham's criteria.
identify differences in bacterial and fungal of the microbial exposome | Month 9
  demonstration of an association between the components of the microbial exposome over an entire year and the response profile to biotherapies used in severe asthma (super-responder vs partial responders), evaluated according to Upham's criteria.
identify differences in bacterial and fungal of the microbial exposome | Month 12
  demonstration of an association between the components of the microbial exposome over an entire year and the response profile to biotherapies used in severe asthma (super-responder vs partial responders), evaluated according to Upham's criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien IMBERT, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - University Hospital, Bordeaux, Bourdeaux
  - University Hospital, Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No